CLINICAL TRIAL: NCT03232645
Title: ELectrical COupling Information From The Rhythmia HDx Mapping System And DireCtSense Technology In The Treatment Of Paroxysmal AtriaL FibrIllation- A Non-RandomiZed, ProspEctive Study
Brief Title: Electrical Coupling Information From The Rhythmia HDx System And DirectSense Technology In Subjects With Paroxysmal Atrial Fibrillation
Acronym: LOCALIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM007
Record Dates: First submitted 2017-07-20; First posted 2017-07-28 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rhythmia HDx and DirectSense technology (Other): Subjects will undergo ablation treatment of the pulmonary veins with the Rhythmia HDx mapping system with DirectSense technology. Subjects indicated for ablation treatment of de-novo PAF will be selected based on the inclusion/exclusion criteria and if deemed to be eligible for participation, will be asked to sign the Informed Consent Form.
  For all enrolled subjects who undergo the ablation procedure, the subjects will be treated with the commercial Rhythmia HDx System with commercially available Software Version 2.0 with DirectSense technology (or any commercially available updates that are released during the course of the study); the IntellaMap Orion mapping catheter and the IntellaNav MiFi OI ablation catheter.
  Interventions: Device: Ablation procedure

INTERVENTIONS:
Device: Ablation procedure — Cathater ablation of pulmonary veins with the Rhythmia HDx mapping system, IntellaMap Orion mapping catheter and IntellaNav Mifi OI ablation catheter

SUMMARY:
The objective of the study is to collect data on the use of the Rhythmia HDx mapping system running commercially available Software Version 2.0 or any future commercially available Software Version with DirectSense technology and the IntellaMap OrionTM mapping catheter in patients indicated for ablation treatment for de-novo Paroxysmal Atrial Fibrillation (PAF). The study will collect specific information to characterize the DirectSense technology in subjects undergoing catheter-based endocardial mapping and ablation for de-novo PAF using a commercial Rhythmia HDx mapping system. The clinical local impedance data will be used in order to generate usage guidance on the DirectSense local impedance feature in the management of de-novo PAF cases requiring Pulmonary Vein Isolation (PVI) and in order to further develop a future lesion indexing feature.

ELIGIBILITY:
Inclusion Criteria:

* • History of recurrent symptomatic PAF with ≥1 episode reported and documented within the 365 days prior to enrollment; PAF is defined as AF episodes that last ≥30 seconds in duration and terminate within 7 days.

  * Refractory or intolerant to at least one Beta Blocker, Calcium Channel Blocker, Class I OR Class III anti-arrhythmic drug (AAD);
  * Eligible for an ablation procedure with the Rhythmia HDx mapping system (software version 2.0 or any future commercially available Software Version), IntellaMap Orion mapping catheter and IntellaNav MiFi OI ablation catheter according to current international and local guidelines (and future revisions) and per physician discretion;
  * Subjects who are willing and capable of providing informed consent;
  * Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center;
  * Age 18 to 80

Exclusion Criteria:

* • Diagnosed with any of the following heart conditions within 90 days (3 months) prior to enrollment:

  1. New York Heart Association (NYHA) Class III or IV
  2. Left ventricular ejection fraction (LVEF) <35%
  3. Left atrial (LA) diameter >5.5 cm
  4. Unstable angina or ongoing myocardial ischemia (OMI)
  5. Transmural myocardial infarction (MI), acute coronary syndrome (ACS), percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery

     * Active systemic infection or sepsis;
     * Undergone any left atrial heart ablation procedure, either surgical or catheter ablation
     * Prosthetic or stenotic valves in the chamber where the intended mapping will occur, or in the path of the catheter access route
     * Subject has a Left Atrial Appendage Closure (LAAC) or Percutaneous Transcatheter Closure of a Patent Foramen Ovale (PFO)
     * Subject has persistent or long-standing persistent atrial fibrillation (AF) ( >1 AF episodes lasting greater than 7 days, with no episodes having lasted greater than 30 days, within the past year)
     * Life expectancy ≤ 6 months per physician judgment
     * Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments; each instance must be brought to the attention of the sponsor to determine eligibility;
     * The subject is unable or not willing to complete follow-up visits and examination for the duration of the study;
     * Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garcia Bolao, MD, Principal Investigator — Clinica Universitaria de Navarra; Bruno Reissmann, MD, Principal Investigator — Universitäres Herzzentrum Hamburg; Armin Luik, MD, Principal Investigator — Stadtisches Klinikum Karlsruhe; Pierre Jais, MD, Principal Investigator — University Hospital, Bordeaux; Moloy Das, MD, Principal Investigator — Freeman Health System; Waqas Ullah, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (6):
- CHU de Bordeaux, Bordeaux, France
- Germany (2):
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Stadtisches Klinikum Karlsruhe, Karlsruhe
- Clinica Universitaria de Navarra, Pamplona, Spain
- United Kingdom (2):
  - Freeman Hospital, Newcastle
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html

REFERENCES:
- [Derived] Garcia-Bolao I, Ramos P, Luik A, S Sulkin M, R Gutbrod S, Oesterlein T, I Laughner J, Richards E, Meyer C, Yue A, Ullah W, Shepherd E, Das M. Local Impedance Drop Predicts Durable Conduction Block in Patients With Paroxysmal Atrial Fibrillation. JACC Clin Electrophysiol. 2022 May;8(5):595-604. doi: 10.1016/j.jacep.2022.01.009. Epub 2022 Feb 23. PMID 35589172

RESULTS

PARTICIPANT FLOW:
Groups:
- Rhythmia HDx and DirectSense Technology: Subjects will undergo ablation treatment of the pulmonary veins with the Rhythmia HDx mapping system with DirectSense technology. Subjects indicated for ablation treatment of de-novo PAF will be selected based on the inclusion/exclusion criteria and if deemed to be eligible for participation, will be asked to sign the Informed Consent Form.
  For all enrolled subjects who undergo the ablation procedure, the subjects will be treated with the commercial Rhythmia HDx System with commercially available Software Version 2.0 with DirectSense technology (or any commercially available updates that are released during the course of the study); the IntellaMap Orion mapping catheter and the IntellaNav MiFi OI ablation catheter.
  Ablation procedure: Cathater ablation of pulmonary veins with the Rhythmia HDx mapping system, IntellaMap Orion mapping catheter and IntellaNav Mifi OI ablation catheter.
  Each subject undergoing PVI will be followed at index procedure, at pre-discharge visit, at the month 3 assessment and at month 4 follow up. The visit at three months after index procedure will include an invasive evaluation with the Rhythmia Mapping system to evaluate residual conduction gaps after PVI.
Period: Overall Study
Arm/Group | Rhythmia HDx and DirectSense Technology
Started | 62
Completed | 58
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Rhythmia HDx and DirectSense Technology: Subjects will undergo ablation treatment of the pulmonary veins with the Rhythmia HDx mapping system with DirectSense technology. Subjects indicated for ablation treatment of de-novo PAF will be selected based on the inclusion/exclusion criteria and if deemed to be eligible for participation, will be asked to sign the Informed Consent Form.
  For all enrolled subjects who undergo the ablation procedure, the subjects will be treated with the commercial Rhythmia HDx System with commercially available Software Version 2.0 with DirectSense technology (or any commercially available updates that are released during the course of the study); the IntellaMap Orion mapping catheter and the IntellaNav MiFi OI ablation catheter.
  Ablation procedure: Catheter ablation of pulmonary veins with the Rhythmia HDx mapping system, IntellaMap Orion mapping catheter and IntellaNav Mifi OI ablation catheter
Arm/Group | Rhythmia HDx and DirectSense Technology
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 62 subjects enrolled, 61 baseline: 1 subject withdrawn consent before baseline
  years
    number analyzed (Participants) | 61
    (all) | 62 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 62 subjects enrolled, 61 baseline: 1 subject withdrawn consent before baseline
  Participants
    number analyzed (Participants) | 61
    Female | 28
    Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19
  France | 1
  Germany | 12
  Spain | 30
Height [Mean (Standard Deviation); unit: cm] — Population: 62 subjects enrolled, 61 baseline: 1 subject withdrawn consent before baseline
  cm
    number analyzed (Participants) | 61
    (all) | 172 (9)
Weight [Mean (Standard Deviation); unit: kg] — Population: 62 subjects enrolled, 61 baseline: 1 subject withdrawn consent before baseline
  kg
    number analyzed (Participants) | 61
    (all) | 80 (12)
Resting Heart Rate [Mean (Standard Deviation); unit: bpm] — Population: 62 subjects enrolled, 61 baseline: 1 subject withdrawn consent before baseline
  bpm
    number analyzed (Participants) | 61
    (all) | 66 (15)
Systolic Blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: 62 subjects enrolled, 61 baseline: 1 subject withdrawn consent before baseline
  mmHg
    number analyzed (Participants) | 61
    (all) | 126 (16)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: 62 subjects enrolled, 61 baseline: 1 subject withdrawn consent before baseline. For one additional subject the data was not collected
  mmHg
    number analyzed (Participants) | 60
    (all) | 72 (9)

OUTCOME MEASURES:

1. Primary Outcome: Local Impedance and Local Impedance Change at Day Zero and PVI Gaps at the Month 3 Assessment
Description: Association between baseline DirectSense data (Local Impedance/Local Impedance change values) per anatomical segment of the Pulmonary Veins at index ablation procedure (Day 0) and the number of ablation gaps per anatomical segment* of the Pulmonary Veins as measured at the month 3 assessment. The outcome is a comparison of local impedance metrics in block versus reconnected segments as assessed at the 3 Month procedure.
  *Each PV pair is divided in 8 segments using tags placed on the left atrium geometry created with the Rhythmia system.
Time Frame: Day 0 and 3 months
Population: 51 subjects were included in the analysis as 7 subjects were removed because the electro-anatomical maps were not technically usable per the specific endpoint analysis.
Measure: Median (Inter-Quartile Range); unit: ohm
Units Other Than Participants: Overall number of Ablations
Arm/Group | Rhythmia HDx and DirectSense Technology
Number analyzed (Participants) | 51
Number analyzed (Overall number of Ablations) | 3872
ohm
  Local Impedance at Baseline in Pulmonary Veins segments where block was achieved | 106.2 [96.6 to 117.4]
  Local Impedance at Baseline in Pulmonary Veins segments where block was not achieved | 101.9 [92.8 to 113.9]
  Local Impedance change in Pulmonary Veins segments where block was achieved | -19.6 [-27.5 to -13]
  Local Impedance change in Pulmonary Veins segments where block was not achieved | -13.9 [-21.5 to -8.8]

2. Secondary Outcome: Local Impedance and Local Impedance Change and PVI Gaps at Day Zero
Description: Acute isolation gaps per anatomical segment* as associated with baseline Local Impedance and Local Impedance change values at first pass encircling during the index ablation procedure (Day 0). The outcome is a comparison of local impedance metrics in block versus reconnected segments as assessed at the index procedure (Day 0).
  *Each PV pair is divided in 8 segments using tags placed on the left atrium geometry created with the Rhythmia system.
Time Frame: Day 0
Population: 55 subjects were included in the analysis as 5 subjects were removed because the electro-anatomical maps were not technically usable per the specific endpoint analysis.
Measure: Median (Inter-Quartile Range); unit: ohm
Units Other Than Participants: Overall number of Ablations
Groups:
- Rhythmia HDx and DirectSense Technology: Subjects will undergo ablation treatment of the pulmonary veins with the Rhythmia HDx mapping system with DirectSense technology. Subjects indicated for ablation treatment of de-novo PAF will be selected based on the inclusion/exclusion criteria and if deemed to be eligible for participation, will be asked to sign the Informed Consent Form.
  For all enrolled subjects who undergo the ablation procedure, the subjects will be treated with the commercial Rhythmia HDx System with commercially available Software Version 2.0 with DirectSense technology (or any commercially available updates that are released during the course of the study); the IntellaMap Orion mapping catheter and the IntellaNav MiFi OI ablation catheter.
  Ablation procedure: Cathater ablation of pulmonary veins with the Rhythmia HDx mapping system, IntellaMap Orion mapping catheter and IntellaNav Mifi OI ablation catheter
Arm/Group | Rhythmia HDx and DirectSense Technology
Number analyzed (Participants) | 55
Number analyzed (Overall number of Ablations) | 3750
ohm
  Local Impedance at Baseline in Pulmonary Veins segments where block was achieved | 107 [97.5 to 118.1]
  Local Impedance at Baseline in Pulmonary Veins segments where block was not achieved | 101.1 [92.5 to 112]
  Local Impedance change in Pulmonary Veins segments where block was achieved | -19.4 [-27.5 to -12.8]
  Local Impedance change in Pulmonary Veins segments where block was not achieved | -10.9 [-18 to -6.6]

3. Secondary Outcome: Number of Gaps at Day Zero
Description: At the index procedure (Day 0), a 20-minute waiting period was required prior to assessing isolation with a left atrium map created with the Rhythmia system. Number and location of gaps for each PV per segment were collected. The outcome is reported as the mean number of gaps per each PV pair.
Time Frame: Day 0
Measure: Mean (Standard Deviation); unit: Number of gaps
Arm/Group | Rhythmia HDx and DirectSense Technology
Number analyzed (Participants) | 60
Number of gaps
  Number of gaps per Left PV pair after initial encircling | 1.4 (1.6)
  Number of gaps per Right PV pair after initial encircling | 1.5 (1.6)

4. Secondary Outcome: Baseline Local Impedance and Local Impedance Change at Day Zero
Description: Average baseline local impedance and local impedance change measured at the index procedure (Day 0) for ablations performed during the first encirclement of the PVs and during the touch ups ablations performed after the 20 minute wait period.
Time Frame: Day 0
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ohm
Units Other Than Participants: Overall number of Ablations
Arm/Group | Rhythmia HDx and DirectSense Technology
Number analyzed (Participants) | 55
Number analyzed (Overall number of Ablations) | 4224
ohm
  Baseline Local Impedance during initial applications | 107.9 (15.9)
  Baseline Local Impedance during touch up applications | 96.1 (13)
  Local Impedance change during initial applications | -19.8 (11.1)
  Local Impedance change during touch up applications | -20.2 (9.5)

5. Secondary Outcome: Maximum Number of Gaps Per PV Segment at Day Zero
Description: At the index procedure (Day 0), a 20-minute waiting period was required prior to assessing isolation with a left atrium map created with the Rhythmia system. Number and location of gaps for each PV per segment were collected.The outcome is reported as the maximum number of gaps identified within segments for each PV pair.
Time Frame: Day 0
Measure: Number; unit: Number of gaps
Arm/Group | Rhythmia HDx and DirectSense Technology
Number analyzed (Participants) | 60
Number of gaps
  Maximum # of gaps observed in a left PV pair segment at index procedure = along appendage/LA ridge | 25
  Maximum # of gaps observed in a right PV pair segment at index procedure = near LA roof | 18

6. Secondary Outcome: Local Impedance in Segments With Maximum Number of Gaps at Day Zero
Description: Local Impedance measured at the index procedure (Day 0) in different anatomical sites of the PV pairs. It is reported the average baseline local impedance in the right and left segments with the maximum number of gaps
Time Frame: Day 0
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ohm
Units Other Than Participants: Overall number of Ablations
Arm/Group | Rhythmia HDx and DirectSense Technology
Number analyzed (Participants) | 55
Number analyzed (Overall number of Ablations) | 3750
ohm
  Average baseline local impedance in left PV segment with maximum gaps = along appendage/LA ridge | 105.2 (13.5)
  Average baseline local impedance in right PV segment with maximum gaps = near LA roof | 105.1 (14.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to end of follow-up: 4 Months.
Description: Reportable Events: All Serious Adverse Events; All Events Leading to Death; All Thromboembolic Events; All Procedure Related AEs; All Rhythmia HDx mapping system, IntellaMap Orion mapping catheter and IntellaNav MiFi OI ablation catheter; Device Related AEs; All Device Deficiencies related to the study devices; Unanticipated Adverse Device Effects/Unanticipated Serious Adverse Device Effects previously not defined in the physicians manuals.
Arm/Group | Rhythmia HDx and DirectSense Technology
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 8/62
Other Adverse Events (participants affected / at risk) | 4/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rhythmia HDx and DirectSense Technology (N=62)
Infection (Surgical and medical procedures) | 2 (2)
Adverse reaction - Neurological (non-TIA, non-stroke) (Surgical and medical procedures) | 1 (1) — Unresponsiveness and Acute Confusion
Stroke (ischemic) (Surgical and medical procedures) | 2 (2)
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pain in the lower stomach, ague, ascites, pleural effusion
Sinus Bradycardia (Cardiac disorders) | 1 (1) — Slow sinus rhythm leading to dizziness
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rhythmia HDx and DirectSense Technology (N=62)
Hemoptosis (Surgical and medical procedures) | 1 (1)
Left Atrial (type II) Flutter (Surgical and medical procedures) | 1 (1) — Atypical Flutter
NSVT (Non Sustained Ventricular Tachycardia) (Surgical and medical procedures) | 1 (1)
Pseudoaneurysm (Surgical and medical procedures) | 1 (1) — Radial Artery Pseudoaneurysm
Visual blurring/disturbances (Surgical and medical procedures) | 1 (1)
Atrial Flutter, not specified (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT03232645/Prot_SAP_000.pdf